CLINICAL TRIAL: NCT04204525
Title: Evidence for Central Sensitization in Patients With Chronic Whiplash Associated Disorders Based on Self-reported Outcomes of Pain (Beliefs), Disability, Central Sensitization, Quantitative Sensory Testing, and Electro-encephalography.
Brief Title: Chronic Whiplash Associated Disorders: Disability, Pain (Beliefs), Central Sensitization and Brain Activity
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other); University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/0850
Record Dates: First submitted 2019-11-20; First posted 2019-12-19 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2019-12

CONDITIONS: Whiplash
Keywords: chronic whiplash associated disorders; central sensitization; electroencephalography; functionality; quality of life; cross-sectional
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic whiplash associated disorders: Male or female, aged between 18 and 65 years. Inclusion: 1) whiplash trauma (at least three months old) and pain since at least 3 months, self-reported mild to severe pain-related disability (score of 5/50 or more on the neck disability index), classified as wad II or wad III on the modified Quebec task force scale; 2) not undertaking exercise 1 day before the experiment; 3) not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state); 4) native dutch speaker and 5) refraining from non-opioid analgesics 48h before the assessments, and refraining from caffeine, alcohol and nicotine 24h before the assessments
  Interventions: Diagnostic Test: Quantitative sensory testing
- Healthy controls: Male or female, aged between 18 and 65 years. Inclusion: 1) no history of whiplash trauma, no pain with a mean pain intensity of more than 2/10 on the visual analogue scale for > 8 consecutive days in the preceding year in the neck-shoulder-arm region 2) painfree at the day of testing 3) native dutch speaker and 4) refraining from non-opioid analgesics 48h before the assessments, and refraining from caffeine, alcohol and nicotine 24h before the assessments.
  Interventions: Diagnostic Test: Quantitative sensory testing

INTERVENTIONS:
Diagnostic Test: Quantitative sensory testing — Electrical detection and pain thresholds will be determined (at the sural nerve of the dominant leg and at the median nerve of both arms) with a constant current electrical stimulator.
  Endogenous pain facilitation will be assessed by a temporal summation paradigm by delivering 20 electrical stimuli at the intensity of the electrical pain threshold.
  Endogenous pain inhibition will be assessed by a conditioned pain modulation paradigm with electrical stimulation as test stimulus and the cold pressor test as conditioning stimulus.
  EEG measurements with be performed with scalp EEG with 32 surface Sn electrodes in a headcap in referential montage following the standard 10-20 recording system.
  A 5 minute resting state measurement will be performed with eyes closed, followed by EEG measurements during the condition pain modulation paradigm to assess the evoked-related potentials.
  Other Names: Electro-encephalography

SUMMARY:
This is a cross-sectional case-control study in which 70 patients with chronic whiplash associated disorders will be recruited and compared to 70 healthy pain-free controls. The primary research question is to determine differences is self-reported functional status, pain, health-related quality of life, psychological correlates, measures of central sensitization, quantitative sensory testing (QST) and quantitative scalp Electroencephalography (EEG) to measure various parameters of brain activation. The secondary research question is to determine whether relationships can be found between the self-reported outcomes on one hand and the QST and EEG on the other hand.

DETAILED DESCRIPTION:
Chronic whiplash associated disorders (CWAD) are frequently occuring conditions with varying degrees of neck pain and disability. They occur usually as a consequence of a motor vehicle accident. Acute whiplash injury has an annual incidence of 200-300 per 100.000 and affects 83% of persons in a traffic collision. Up to 50% of WAD patients do not fully recover, and up to 25% continue to have moderate to severe pain-related disabilities. The consequent pain and disability give rise to substantial socioeconomic cost. In Europe, the annual cost of WAD was estimated to be 12 billion euro.

Chronic neck pain, as observed in CWAD, is often incompletely responsive to available therapies. Due to the current lack of knowledge concerning the underlying factors responsible for the maintenance of these chronic pain conditions, there is no consensus on dedicated and specific therapy approaches for CWAD, resulting in a treatment gap in this condition. The chronicity and severeness of the disorders has led to paradigm shifts in the reasoning about chronic pain from seeing it as a symptom towards as a disease. Neuroimaging has provided evidence that chronic pain is a multidimensional process affecting sensory and emotional processing based on an altered state of the central nervous system in the form of central sensitization (CS). This sensitization results from an increased responsiveness to a variety of stimuli and expresses itself in the form of hyperalgesia, allodynia, referred pain, and ultimately in chronic widespread pain. Changes in both structural and functional brain activity and connectivity over time contribute to an augmentation of pain perception, by an enhanced pain facilitation and defective inhibition of nociceptive signals. It remains however debated whether CS is present as a pathophysiological feature in CWAD.

In this project we hypothesize that CS is one of the main features of the pathophysiology of CWAD, and that relationships occur between QST and EEG on one hand, and self-reported pain, disability, quality of life, psychological correlates and central sensitization on the other hand.

Therefore, 70 patients with CWAD and 70 (gender and age) matched healthy controls will be invited to fill out questionnaires, perform a QST protocol and EEG measurements.

The questionnaires will be filled out online during the two weeks before the determined testing moment and will consist of the Neck Disability Index, the Short Form Health Survey-36 items, a 0-10 Numeric Rating Scale for pain, the Central Sensitization Inventory, the Dutch version of the Pain Catastrophizing Scale, the Impact of Event Scale revised, the Pain anxiety symptoms scale (PASS-20), the patient specific complaints questionnaire (PSK), the Dolour neuropathic 4 (DN4) and the Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS). Dutch versions of all questionnaires will be used.

During the testing moment, a QST protocol will be combined with EEG assessment. Electrical detection and electrical pain thresholds will be determined with a constant current electrical stimulator (DS7A Digitimer). Determination of the electrical detection and electrical pain threshold with the electrical stimulator will be performed at the sural nerve of the dominant leg and at the median nerve of both arms. Endogenous pain facilitation will be assessed by a temporal summation paradigm by delivering 20 electrical stimuli at the intensity of the electrical pain threshold.

Endogenous pain inhibition will be assessed by a conditioned pain modulation paradigm with electrical stimulation as test stimulus and the cold pressor test (immersion of the hand up to the wrist in cold water of 12°C) as conditioning stimulus.

EEG measurements with be performed with scalp EEG (Eego Sports, Ant neuro) with 32 surface Sn electrodes in a headcap in referential montage following the standard 10-20 recording system. Participants will be seated in a comfortable chair in a quiet room.

A 5 minute resting state measurement will be performed with eyes closed, followed by EEG measurements during the condition pain modulation paradigm.

ELIGIBILITY:
Patients with chronic WAD (n=70), male or female, aged between 18 and 65 years, will be recruited.

The patients should meet the following inclusion criteria: 1) a whiplash trauma which is at least three months old and causes pain since at least 3 months, with self-reported mild to severe pain-related disability, established by a score of 5 or more of a maximum of 50 on the neck disability index, patients classified as wad II or wad III on the modified Quebec task force scale; 2) not undertaking exercise 1 day before the experiment; 3) not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state); 4) native dutch speaker and 5) refraining from non-opioid analgesics 48h before the assessments, and refraining from caffeine, alcohol and nicotine 24h before the assessments.

Exclusion criteria:

Neuropathic pain; being pregnant or having given birth in the preceding year; chronic fatigue syndrome, fibromyalgia, cardiovascular disorders, endocrinological disorders, rheumatic and psychiatric disorders, epilepsy, history of specific spinal surgery (i.e. surgery for spinal stenosis); history of neck or shoulder surgery in the past 3 years and loss of consciousness during/after the trauma.

Healthy pain-free persons (n=70), male or female, aged between 18 and 65 years, will be recruited. The healthy pain-free persons will serve as a control group and should meet the following inclusion criteria: 1) no history of whiplash trauma, no pain experience with a mean pain intensity of more than 2 out of 10 on the visual analogue scale for more than 8 consecutive days in the preceding year in the neck-shoulder-arm region 2) painfree at the day of testing (vas < 2/10) 3) native dutch speaker and 4) refraining from non-opioid analgesics 48h before the assessments (experimental measures baseline), and refraining from caffeine, alcohol and nicotine 24h before the assessments (experimental measures baseline).

Exclusion criteria:

being pregnant or having given birth in the preceding year; chronic fatigue syndrome, fibromyalgia, cardiovascular disorders, endocrinological or neurological disorders, rheumatic and psychiatric disorders, epilepsy, history of neck-shoulder surgery.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic whiplash associated disorders will be compared to healthy controls
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Self-reported functional status or disability | Single assessment, within 2 weeks before test moment
  The Dutch version of the Neck Disability Index (questionnaire)
Self-reported health-related quality of life | Single assessment, within 2 weeks before test moment
  The Dutch version of the Short Form Health Survey-36 items (questionnaire)
Self-reported pain assessment | Single assessment, at test moment
  A 0-10 Numeric Rating Scale for pain (questionnaire). Patients fill out the Numeric Rating Scale (0 no pain - 10 worst pain imaginable) for their perceived neck pain.
Self-reported central sensitization symptoms | Single assessment, within 2 weeks before test moment
  The Dutch version of the Central Sensitization Inventory (questionnaire)
Electrical detection and electrical pain thresholds with a constant current electrical stimulator (DS7A Digitimer) | Single assessment, during single test moment (duration: approximately 20min), date of test moment will be determined based on the availability of the subject.
  Determination of the electrical detection and electrical pain threshold with the electrical stimulator will be performed at the sural nerve of the dominant leg and at the median nerve of the arms.
Endogenous pain facilitation assessed by a temporal summation paradigm | Single assessment, during single test moment (duration: approximately 10min), date of test moment will be determined based on the availability of the subject.
  Temporal summation of electrical pain will be assessed by delivering 20 electrical stimuli at the intensity of the electrical pain threshold.
Endogenous pain inhibition assessed by a conditioned pain modulation paradigm | Single assessment,during single test moment (duration: approximately 10min), date of test moment will be determined based on the availability of the subject.
  Conditioned pain modulation will be tested with electrical stimulation as test stimulus and the cold pressor test (immersion the hand up to the wrist in cold water of 12°C) as conditioning stimulus.
Resting state brain activity | Single assessment, during single test moment (duration: approximately 5min), date of test moment will be determined based on the availability of the subject.
  Quantitative Electroencephalography (QEEG) will be recorded from 32 Sn surface electrodes using an electrode cap during 5 minutes of sitting on a chair with eyes closed. Spectral power will be analyzed.
Event-related potentials | Single assessment, during single test moment (duration: approximately 20min), date of test moment will be determined based on the availability of the subject.
  Quantitative Electroencephalography (QEEG) will be recorded from 32 Sn surface electrodes using an electrode cap during the conditioned pain modulation paradigm. Latency and amplitude of the event-related potentials will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Coppieters, Study Director — University Ghent; Jo Nijs, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Ghent university, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pinheiro ES, de Queiros FC, Montoya P, Santos CL, do Nascimento MA, Ito CH, Silva M, Nunes Santos DB, Benevides S, Miranda JG, Sa KN, Baptista AF. Electroencephalographic Patterns in Chronic Pain: A Systematic Review of the Literature. PLoS One. 2016 Feb 25;11(2):e0149085. doi: 10.1371/journal.pone.0149085. eCollection 2016. PMID 26914356
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Paul L. Evidence for central sensitization in chronic whiplash: a systematic literature review. Eur J Pain. 2013 Mar;17(3):299-312. doi: 10.1002/j.1532-2149.2012.00193.x. Epub 2012 Sep 25. PMID 23008191
- [Derived] Lenoir D, Willaert W, Ickmans K, Bernaers L, Nijs J, Malfliet A, Danneels L, Leysen L, De Pauw R, Cagnie B, Coppieters I, Meeus M. Are Reports of Pain, Disability, Quality of Life, Psychological Factors, and Central Sensitization Related to Outcomes of Quantitative Sensory Testing in Patients Suffering From Chronic Whiplash Associated Disorders? Clin J Pain. 2021 Dec 22;38(3):159-172. doi: 10.1097/AJP.0000000000001013. PMID 34939972